CLINICAL TRIAL: NCT03747679
Title: A SINGLE-BLIND, RANDOMIZED, MULTIPLE-PERIOD STUDY IN HEALTHY ADULT VOLUNTEERS TO INVESTIGATE THE PALATABILITY OF PROTOTYPE AGE APPROPRIATE ORAL FORMULATIONS OF BOSUTINIB FOR PEDIATRIC USE
Brief Title: Palatability (Taste) of Oral Formulations of Bosutinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: B1871057; 2018-002346-37 (EudraCT Number); BCHILD TASTE (Other: Alias Study Number)
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: CML
Keywords: CML; palatability; taste; pediatric formulation
MeSH Terms: interventions — bosutinib

STUDY DESIGN:
Intervention Model Description: This will be a single-blind, randomized, multiple-period (dosing over 4 days) study in healthy male and/or female participants. Approximately 8 participants will assess the sensory attributes of each of the formulation options using Bosutinib Taste Assessment Questionnaire
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- A- Bosutinib in water (Experimental): 200 Mg of bosutinib (50 mg capsule x4) in Water solution
  Interventions: Drug: 200 Mg capsules of bosutinib in Water solution
- B- bosutinib in sorbitol (Experimental): 200 Mg of bosutinib sorbitol base in water solution
  Interventions: Drug: bosunitib sorbitol
- C- - bosutinib mannitol (Experimental): 200 Mg of bosutinib powder mannitol base in water solution
  Interventions: Drug: Bosutinib Mannitol
- D - bosutinib in mannitol low sweet (Experimental): 200 Mg of bosutinib mannitol low sweet solution
  Interventions: Drug: bosutinib in mannitol low sweet
- E- - bosutinib in mannitol high sweet (Experimental): 200 Mg of bosutinib High % sweet mannitol solution
  Interventions: Drug: bosutinib in mannitol high sweet
- F- - bosutinib low flavour (Experimental): Taste assessment of 200 Mg of bosutinib low % Flavour
  Interventions: Drug: bosutinib taste low flavour
- G- bosutinib high flavour (Experimental): Taste assessment of 200 Mg of bosutinib high percentage of flavor in water
  Interventions: Drug: bosutinib high flavour
- H- - bosutinib capsules in low sweet (Experimental): Taste assessment of 200 Mg of bosutinib (50 mg x4 capsules) low % sweet
  Interventions: Drug: Bosutinib capsules in low sweet
- I - bosutinib capsules high sweet (Experimental): 200 Mg of bosutinib (4 X 50 mg capsules)in high % sweetener
  Interventions: Drug: bosutinib capsules high sweet
- J- - bosutinib capsules low flavour (Experimental): Taste assessment of 200 Mg of bosutinib (50 mg X4 capsules) in Low % flavour Water solution
  Interventions: Drug: bosutinib capsules low flavour
- K - bosutinib capsules high flavour (Experimental): Taste assessment of 200 Mg of bosutinib (50 mg X 4 capsules) in high % flavour
  Interventions: Drug: bosutinib capsules high flavour
- L - bosutinib capsules applesauce (Experimental): 200 Mg of bosutinib (50 mg x 4 capsules) in applesauce
  Interventions: Drug: bosutinib capsules in applesauce
- M - bosutinib capsules full fat yougurt (Experimental): 200 Mg of bosutinib (50 mg x 4 capsules) in full fat yogurt
  Interventions: Drug: Bosutinib capsules in yogurt
- N - bosutinib capsules in water (retest) (Experimental): 200 Mg of bosutinib (50 mg x 4 capsules) in Water (retest)
  Interventions: Drug: bosutinib capsules in water

INTERVENTIONS:
Drug: 200 Mg capsules of bosutinib in Water solution — 200 mg (4X50) Capsules in water
  Arms: A- Bosutinib in water
Drug: bosunitib sorbitol — 200 Mg of bosutinib sorbitol solution
  Arms: B- bosutinib in sorbitol
Drug: Bosutinib Mannitol — Bosutinib mannitol solution
  Arms: C- - bosutinib mannitol
Drug: bosutinib in mannitol low sweet — bosutinib in mannitol solution low sweet
  Arms: D - bosutinib in mannitol low sweet
Drug: bosutinib in mannitol high sweet — bosutinib in mannitol high sweet
  Arms: E- - bosutinib in mannitol high sweet
Drug: bosutinib taste low flavour — bosutinib solution low flavour
  Arms: F- - bosutinib low flavour
Drug: bosutinib high flavour — bosutinib solution high flavour
  Arms: G- bosutinib high flavour
Drug: bosutinib capsules in applesauce — Bosutinib capsules in applesauce
  Arms: L - bosutinib capsules applesauce
Drug: Bosutinib capsules in yogurt — bosutinib capsules in yogurt
  Arms: M - bosutinib capsules full fat yougurt
Drug: bosutinib capsules in water — sham comparator, bosutinb in water retest
  Arms: N - bosutinib capsules in water (retest)
Drug: Bosutinib capsules in low sweet — bosutinib capsules in low sweet
  Arms: H- - bosutinib capsules in low sweet
Drug: bosutinib capsules high sweet — Bosutinib capsules high sweet
  Arms: I - bosutinib capsules high sweet
Drug: bosutinib capsules low flavour — Bosutinib capsules low flavour
  Arms: J- - bosutinib capsules low flavour
Drug: bosutinib capsules high flavour — bosutinib capsules in high flavour
  Arms: K - bosutinib capsules high flavour

SUMMARY:
Healthy Adult Volunteer Taste Study of Oral Formulations of Bosutinib for Pediatric Use. This will be a single-blind, randomized, multiple-period (dosing over 4 days) study in healthy male and/or female participants. Approximately 8 participants will assess the sensory attributes of different powder for oral suspension (POS) formulations.

DETAILED DESCRIPTION:
Taste evaluations for the formulations (Formulations A to N) in Sessions 1 to 4 each contains 4 periods. All the planned formulations in this study will have a bosutinib amount equal to 200 mg in each taste assessment. Session 1 consists of bosutinib POS, sorbitol base in water (A); bosutinib POS, mannitol base in water (B); and bosutinib capsules to be opened into water (C). Session 2 consists of bosutinib POS, mannitol base in low % (D) and in high % (E) sodium saccharine sweetener vehicles, respectively; bosutinib POS, mannitol base in low % (F) and high % (G) strawberry flavour vehicles, respectively. Session 3 consists of bosutinib capsules to be opened into low % (H) and high % (I) sodium saccharine sweetener vehicles, respectively; bosutinib capsules to be opened into low % (J) and high % (K) strawberry flavour vehicles, respectively. Session 4 consists of bosutinib capsules opened onto apple sauce (L); bosutinib capsules opened onto full fat natural yoghurt (M); and bosutinib capsules to be opened into water (N). Participants will be assigned to one of the treatment sequences available for each session. Except at session 4 for treatments L and M, each formulation will be presented to the participants in a blinded fashion.

Participants will be required to not swallow, rather to only swish the bosutinib containing liquid in their mouths for approximately 10 seconds, after which the liquid will be spat out. Each participant will record the sensory attributes at timed intervals of 0 (immediately after dosing), 5, 10 and 20 minutes after spitting using a Bosutinib Taste Assessment Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Age and Sex:

1. Female participants of non-childbearing potential and/or male participants able to father children must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD).

   -Refer to Appendix 4 for reproductive criteria for male (Section 10.4.1) and female (Section 10.4.2) participants.

   Type of Participant and Disease Characteristics:
2. Male and female participants who are overtly healthy as determined by medical evaluation including a detailed medical history, limited physical examination, including blood pressure (BP) and pulse rate measurement, or clinical laboratory tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

   Weight:
4. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >45 kg (99 lbs).

   Informed Consent:
5. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria:

Medical Conditions:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. A history of hypersensitivity to the active compounds or to any inactive ingredients (excipients) contained in the formulations.
3. Participants with conditions that affect their ability to taste - ie, dysgeusia, respiratory infection, cold, etc.
4. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C antibody (HCVAb). As an exception, a positive hepatitis B surface antibody (HBsAb) as a result of participant vaccination is permissible.
5. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

   Prior/Concomitant Therapy:
6. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product. (Refer to Section 6.5 for additional details).

   Prior/Concurrent Clinical Study Experience:
7. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product used in this study (whichever is longer).

   Diagnostic Assessments:
8. A positive urine drug test.
9. Use of tobacco-containing products.
10. Screening supine blood pressure (BP) 140 mm Hg (systolic) or 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is 140 mm Hg (systolic) or 90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
11. Baseline 12 lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline corrected QT (QTc) interval >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
12. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level 1.5 × upper limit of normal (ULN);
    * Total bilirubin level 1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ULN.

    Other Exclusions:
13. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of consuming 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
14. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
15. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
16. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.
17. Male participants with partners currently pregnant; male participants able to father children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product or longer based upon the compound's half-life characteristics.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib in Water) | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib sorbitol) | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib mannitol) | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib mannitol low sweet) | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use(Bosutinib mannitol high sweet) | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib mannitol in low flavour strawberry) | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib mannitol high flavour strawberry) | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib 50 mg capsules X4) low sweet | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib 50 mg capsules X4) high sweet | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib 50 mg capsules X4) low flavour | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib 50 mg capsules X4) high flavour | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib 50 mg capsules X4) applesauce | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (bosutinib 4 capsules 50 mg bosutinib in yogurt | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib
Taste evaluation using Bosutinib Taste Assessment Questionnaire toward formulation for pediatric use (Bosutinib 50 mg capsules X4 in water retest) | baseline to one month
  This study will enable the selection of the commercial formulation for pediatric use of bosutinib

SECONDARY OUTCOMES:
Number or treatment emergent treatment related adverse events following oral administration of bosutinib solution bosutinib 200 mg sorbitol | Baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number or treatment emergent treatment related adverse events following oral administration of 200 mg bosutinib powder mannitol solution | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number of patients with treatment emergent treatment related adverse events bosutinib 50 mg x4 capsules in water | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number of patients with treatment emergent treatment related adverse events bosutinib 200 mg mannitol low sweet | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
number of patients with treatment emergent or treatment related adverse events bosutinib 200 mg mannitol high sweet | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
number of patients with treatment emergent treatment related adverse events bosutinib 200 mg mannitol high flavour (strawberry) | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number or treatment emergent treatment related adverse events following oral administration of bosutinib 200 mg solution mannitol low flavour | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number or treatment emergent treatment related adverse events following oral administration of bosutinib solution 50 mg x 4 capsules high sweet | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number or treatment emergent treatment related adverse events following oral administration of bosutinib solution capsules 4 x 50mg low flavour | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number or treatment emergent treatment related adverse events following oral administration of bosutinib solution capsules 50 mg X4 high flavour | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number or treatment emergent treatment related adverse events following oral administration of bosutinib solution capsules 4 x 50 mg applesauce | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number or treatment emergent treatment related adverse events following oral administration of bosutinib solution capsules 50 mg x4 in yogurt | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number of treatment emergent treatment related adverse events following oral administration of 4 X50 mg capsules bosutinib low sweet solution | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number of treatment emergent treatment related adverse events following oral administration of bosutinib 50 mg capsules x4 in water (retest) | baseline to one month
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Bosutinib was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1871057